CLINICAL TRIAL: NCT07141706
Title: A Phase 1a/1b, Multicenter, Open-Label, First-in-Human Study to Assess the Safety, Tolerability, Pharmacokinetics, and Preliminary Antitumor Activity of DB-1317 in Participants With Selected Advanced/Metastatic Solid Tumors
Brief Title: A Study of DB-1317 in Selected Advanced/Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: DualityBio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DB-1317-101
Record Dates: First submitted 2025-08-18; First posted 2025-08-26 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Advanced/Metastatic Solid Tumors
Keywords: ADAM9; Solid tumor; DB-1317

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- DB-1317 Dose Level 1 (Experimental): Enrolled Subjects will receive a single-dose of DB-1317 at Dose Level 1 on Day 1 of each cycle Q3W
  Interventions: Drug: DB-1317
- DB-1317 Dose Level 2 (Experimental): Enrolled Subjects will receive a single-dose of DB-1317 at Dose Level 2 on Day 1 of each cycle Q3W
  Interventions: Drug: DB-1317
- DB-1317 Dose Level 3 (Experimental): Enrolled Subjects will receive a single-dose of DB-1317 at Dose Level 3 on Day 1 of each cycle Q3W
  Interventions: Drug: DB-1317
- DB-1317 Dose Level 4 (Experimental): Enrolled Subjects will receive a single-dose of DB-1317 at Dose Level 4 on Day 1 of each cycle Q3W
  Interventions: Drug: DB-1317
- DB-1317 Dose Level 5 (Experimental): Enrolled Subjects will receive a single-dose of DB-1317 at Dose Level 5 on Day 1 of each cycle Q3W
  Interventions: Drug: DB-1317
- DB-1317 Dose Expansion 1 (Experimental): Subjects with advanced/unresectable, or metastatic Gastric cancer (GC) who have progressed on or after standard systemic treatments, a 21-day treatment cycle (i.e., once every 3 weeks) via intravenous infusion will be used for DB-1317
  Interventions: Drug: DB-1317
- DB-1317 Dose Expansion 2 (Experimental): Subjects with advanced/unresectable, or metastatic colorectal cancer (CRC) who have progressed on or after standard systemic treatments, a 21-day treatment cycle (i.e., once every 3 weeks) via intravenous infusion will be used for DB-1317
  Interventions: Drug: DB-1317
- DB-1317 Dose Expansion 3 (Experimental): Subjects with advanced/unresectable, or metastatic pancreatic ductal adenocarcinoma (PDAC) who have progressed on or after standard systemic treatments, a 21-day treatment cycle (i.e., once every 3 weeks) via intravenous infusion will be used for DB-1317
  Interventions: Drug: DB-1317

INTERVENTIONS:
Drug: DB-1317 — Administered I.V.

SUMMARY:
This is a multicenter, open-label, multiple-dose, FIH Phase 1a/1b study. Phase 1a adopts an accelerated titration design and a BOIN design to identify the MTD or MAD of DB-1317; Phase 1b includes up to 3 randomized dose expansion cohorts to further evaluate the safety, tolerability and preliminary efficacy of DB-1317 in selected solid tumors and to identify optimal RP2D.

DETAILED DESCRIPTION:
Phase 1a (Dose Escalation and Backfilling)

Approximately 5 increasing dose levels of DB-1317 dosing every 3 weeks (Q3W) will be evaluated using an accelerated titration design at the first dose level, followed by a BOIN design at subsequent dose levels with the oversight of a Safety Monitoring Committee (SMC). For safety reasons, in any dose level of the dose escalation where a number of participants ≥ 2, a staggered dosing is required. The second participant in each dose level should start dosing no sooner than at least 24 hours after the initial dosing of the first participant. If no safety concerns arise during these 24 hours, the remaining participants can be enrolled into the same dose level with no additional staggering required. Each dose level will be subject to the DLT assessment. After completing the 21-day DLT observation period (Cycle 1), participants will continue to the next treatment cycle and receive DB-1317 on Day 1 of each cycle in the same dose level cohort. Participants who complete the DLT observation period are not allowed to switch to a higher dose level (i.e., intra-participant escalation is not allowed) unless it is deemed necessary and strongly recommended by the investigator with a written approval by the Sponsor.

Phase 1b (Dose Expansion)

Upon completion of the Phase 1a dose escalation, following determination of MTD or MAD, and at the Sponsor's discretion, -one randomized expansion cohort and two single arm expansion cohorts will be opened each enrolling one of the selected solid tumor types, if preliminary anti-tumor activities in these tumor types are observed in Phase 1a part. GC is the tumor type pre-selected for the randomized expansion cohort CRC and PDAC are the two tumor types pre-selected for the single arm expansion cohorts based on ADAM9 expressing data, in vivo anti-tumor activities in non-clinical tumor models, and consideration of unmet medical needs. The final selection of tumor type(s) to be enrolled in the Phase 1b cohorts will be determined by Sponsor based on emerging data from Phase 1a part. Approximately -80 participants will be enrolled in the randomized expansion cohort and randomly assigned in a 1:1 ratio to two dose levels (approximately 40 each) . Approximately 40 participants will be enrolled in each single arm expansion cohort at a selected dose level, and 160 participants will be enrolled in Phase 1b. Dose levels used in Phase 1b part will be determined by Sponsor and SMC based on Phase 1a data. Based on new emerging data from the study, Sponsor may explore other randomized cohorts with other tumor types.

ELIGIBILITY:
Key Inclusion Criteria:

1. Male or female adults
2. Unresectable advanced or metastatic selected solid tumors that have relapsed or progressed on or after standard systemic treatments.
3. Only applicable to backfilling participants in Phase 1a and participants in Phase 1b: At least one measurable lesion as assessed by the investigator according to RECIST version 1.1 criteria. Participants with non-measurable disease are allowed for CRPC participants.
4. Has a life expectancy of ≥ 3 months.
5. Has an ECOG PS of 0-1.
6. Has LVEF ≥ 50% within 28 days before enrollment.
7. Is willing to provide pre-existing resected tumor samples or undergo fresh tumor biopsy for the measurement of ADAM9 expression level and other biomarkers if no contra-indication.
8. Male and female participants of reproductive/childbearing potential must agree to use adequate contraceptive methods

Key Exclusion Criteria:

1. Prior treatment with ADAM9 targeted therapy.
2. Prior treatment with antibody-drug conjugate with topoisomerase I inhibitor.
3. Has a medical history of symptomatic congestive heart failure or serious cardiac arrhythmia requiring treatment.
4. Has a medical history of myocardial infarction or unstable angina within 6 months before enrollment.
5. Has any clinically important abnormalities in rhythm, conduction or morphology of resting ECG
6. Has an average of Fredericia's formula-QT corrected interval (QTcF) prolongation to > 470 ms in males and females
7. Has a history of (non-infectious) ILD/pneumonitis
8. Has a lung-specific intercurrent clinically significant illness
9. Has an uncontrolled infection requiring intravenous injection of antibiotics, antivirals, or antifungals.
10. Known human immunodeficiency virus (HIV) infection;Chronic, active, or uncontrolled hepatitis B;
11. Known chronic, active, or uncontrolled hepatitis C
12. Has clinically significant corneal disease.
13. Has clinically active brain metastases
14. Has unresolved toxicities from previous anticancer therapy Concurrent malignancy < 3 years.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 233 (Estimated)
Dates: Start 2025-09-23 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Phase 1a: Percentage of Participants with Dose-Limiting Toxicities (DLTs) as assessed by CTCAE v5.0. Percentage of participants in Part 1 with DLTs | up to 21 days after Cycle 1 Day 1
  Percentage of participants in Phase 1a with DLTs
Phase 1a: Percentage of Participants with Treatment Emergent Adverse Events (TEAEs) as assessed by CTCAE v5.0. | Up to follow-up period, approximately 1 year post-treatment
  Percentage of participants with TEAEs in Phase 1a graded according to NCI CTCAE v5.0
Phase 1a: Percentage of Participants with Serious Adverse Events (SAEs) as assessed by CTCAE v5.0. | Up to follow-up period, approximately 1 year post-treatment
  Percentage of Participants with SAEs in Phase 1a graded according to NCI CTCAE v5.0
Maximum Tolerated Dose (MTD) of DB-1317 | Up to the completion of Phase 1a (assessed up to 12 months)
  MTD on the data collected during Phase 1a
Recommended Phase 1b Dose (RP2D) of DB-1317 | Up to the completion of Phase 1a (assessed up to 12 months)
  RP2D of DB-1317 based on the data collected during Phase 1a
Phase 1b: Percentage of Participants with Treatment Emergent adverse events (TEAEs) as assessed by CTCAE v5.0. | Up to follow-up period, approximately 1 year post-treatment
  Percentage of participants with TEAEs in Phase 1b graded according to NCI CTCAE v5.0
Phase 1b: Percentage of participants with Serious Adverse Events (SAEs) as assessed by CTCAE v5.0. | Up to follow-up period, approximately 1 year post-treatment
  Percentage of participants with SAEs in Phase 1b graded according to NCI CTCAE v5.0
Phase 1b: Objective Response Rate (ORR) as determined by investigator | Up to follow-up period, approximately 1 year post-treatment
  Phase 1b: Objective Response Rate (ORR) as determined by investigator per RECIST 1.1 in non-CRPC. The percentage of participants who had a best response rating of CR and PR, for Part 2 only which was maintained ≥4 weeks
Phase 1b: duration of response (DoR) | Up to follow-up period, approximately 1 year post-treatment
  DoR will be determined from tumor assessments by investigator per response evaluation criteria in solid tumors version 1.1 (RECIST v1.1)
Phase 1b: disease-control rate (DCR) | Up to follow-up period, approximately 1 year post-treatment
  DCR will be determined from tumor assessments by investigator per response
Phase 1b: Time to Response (TTR) | Up to follow-up period, approximately 1 year post-treatment
  TTR will be determined from tumor assessments by investigator per response

SECONDARY OUTCOMES:
Phase 1a: Objective response rate (ORR) | Up to follow-up period, approximately 1 year post-treatment
  ORR will be determined from tumor assessments by investigator per response evaluation criteria in solid tumors version 1.1 (RECIST v1.1)
Phase 1a: duration of response (DoR) | Up to follow-up period, approximately 1 year post-treatment
  DoR will be determined from tumor assessments by investigator per response evaluation criteria in solid tumors version 1.1 (RECIST v1.1)
Phase 1a: disease-control rate (DCR) | Up to follow-up period, approximately 1 year post-treatment
  DCR will be determined from tumor assessments by investigator per response evaluation criteria in solid tumors version 1.1 (RECIST v1.1)
Phase 1a: Time to Response (TTR) | Up to follow-up period, approximately 1 year post-treatment
  TTR will be determined from tumor assessments by investigator per response evaluation TTR criteria in solid tumors version 1.1 (RECIST v1.1)
Phase 1a & Phase 1b: Progression Free Survival (PFS) | Up to follow-up period, approximately 1 year post-treatment
  PFS will be determined from tumor assessments by investigator per response evaluation PFS criteria in solid tumors version 1.1 (RECIST v1.1)
Phase 1a & Phase 1b: Overall Survival (OS) | From date of first dose until the date of death or lost to follow up, approximately 1 year post-treatment
  OS is defined as the time from date of first dose to the date of death.
Phase 1a: Prostate-specific antigen (PSA) | From date of first dose until the date of first PSA progression, approximately 1 year post-treatment
  Time to PSA progression, PSA50 response rate and PSA90 response rate, duration of PSA response in CRPC subjects.
Phase 1a & Phase 1b: Pharmacokinetic-AUC | within 3 cycles (each cycle is 21 days)
  Area under the concentration-time curve from time 0 to infinity of DB-1317 ADC, total anti-Adam 9 antibody, and unconjugated P1003
Phase 1a & Phase 1b: Pharmacokinetic-Cmax | within 3 cycles (each cycle is 21 days)
  Maximum observed plasma concentration (Cmax) of DB-1317 ADC, total anti-Adam 9 antibody, and unconjugated P1003
Phase 1a & Phase 1b: Pharmacokinetic-Tmax | within 3 cycles (each cycle is 21 days)
  Time to Cmax of DB-1317 ADC, total anti-Adam 9 antibody, and unconjugated P1003
Phase 1a & Phase 1b: Pharmacokinetic-Cthrough | within 6 cycles (each cycle is 21 days)
  Trough concentration
Phase 1a & Phase 1b: Anti-drug antibody (ADA) prevalence | Up to follow-up period, approximately 1 year post-treatment
  Percentage of participants who are ADA positive at any point
Phase 1a & Phase 1b: ADA incidence | Up to follow-up period, approximately 1 year post-treatment
  Percentage of participants having treatment-emergent ADA

CONTACTS AND LOCATIONS:
Overall Officials: Lily Hu, Study Director — DualityBio Inc.
Locations (4):
- United States (3):
  - USA02-0, Houston, Texas
  - USA03-0, San Antonio, Texas
  - USA01, Fairfax, Virginia
- AUS01-0, Randwick, New South Wales, Australia